CLINICAL TRIAL: NCT02198248
Title: Low-dose Glucocorticoids Plus Rituximab Versus High-dose Glucocorticoids Plus Rituximab for Remission Induction in ANCA-associated Vasculitis; a Multicentre, Open Label, Randomised Control Trial
Brief Title: Low-dose Glucocorticoid Vasculitis Induction Study
Acronym: LoVAS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chiba University (Other)
Responsible Party: Principal Investigator, Shunsuke Furuta, Associate Professor, Chiba University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G25051; UMIN000014222 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2014-07-18; First posted 2014-07-23 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Microscopic Polyangiitis; Wegener Granulomatosis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Microscopic Polyangiitis; Granulomatosis with Polyangiitis | interventions — Rituximab; Glucocorticoids; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-dose glucocorticoid (Experimental): Prednisolone will be commenced with dose of 0.5mg/kg/day and will be tapered and off within 6 months. If a patient fails to achieve BVAS=0, an investigator can postpone the procedure of stopping prednisolone (prednisolone 5mg/day x 2 weeks, 4mg/day x 2 weeks, 3mg/day x 4 weeks, 2mg/day x 4 weeks, 1mg/day x 4 weeks, then off prednisolone). Once starting the procedure, prednisolone must be off after 16 weeks. Patients will also receive rituximab (375mg/m2/w x4).
  After achieving remission, patients will be receive rituximab (1g/body or 0.5g/bodyx2) every 6 months as remission maintenance therapy.
  Interventions: Drug: Rituximab; Drug: Glucocorticoids
- High-dose glucocorticoid (Active Comparator): Prednisolone will be commenced with dose of 1.0mg/kg/day and will be tapered to 10mg/day within 6 months. Patients will also receive rituximab (375mg/m2/w x4).
  After achieving remission, patients will be receive rituximab (1g/body or 0.5g/bodyx2) every 6 months as remission maintenance therapy. There's no limitation by the protocol regarding further prednisolone tapering.
  Interventions: Drug: Rituximab; Drug: Glucocorticoids

INTERVENTIONS:
Drug: Rituximab — Patients will be administered rituximab (375mg/m2/w x4 infusions) for reducing glucocorticoid dose in remission induction phase.
  Other Names: Rituxan
Drug: Glucocorticoids — "Low-dose" group commenced 0.5mg/kg/day, then taper and stop within 6 months following pre-defined schedule.
  "High-dose" group commenced 1.0mg/kg/day, then taper to 10mg/day within 6 months following pre-defined schedule.
  Other Names: Predonine; Prednisolone

SUMMARY:
Previous reports suggested conventional immunosuppressants such as cyclophosphamide could not reduce glucocorticoid dose in remission induction in ANCA-associated vasculitis because of lower remission rate and higher relapse rate. However those reports didn't include rituximab.

B cell depletion therapy by rituximab is a new strategy for remission induction in ANCA-associated vasculitis. The RAVE and RITUXVAS trial (NEJM 2010, both) showed high-dose glucocorticoid plus rituximab had roughly the same efficacy and safety as high-dose glucocorticoid plus IV-cyclophosphamide. In addition, recent retrospective observational studies reported low-dose glucocorticoid plus rituximab led to re-induction in severe relapsing ANCA-associated vasculitis.

Thus, the investigators aim to investigate whether rituximab can reduce glucocorticoid dose in induction remission in ANCA-associated vasculitis (to show non-inferiority for efficacy between low-dose and high-dose glucocorticoid plus rituximab). Participants will be randomised to the "low-dose glucocorticoid plus rituximab" or the high-dose glucocorticoid plus rituximab" groups. Primary endpoint is proportion of remission at 6 months, then data regarding relapse and long-term safety will be collected until 24 months.

The study has been designed by the principal and coordinating investigators. It will include 140 participants from 18 hospitals in Japan. It is funded by Chiba University Hospital and Chiba East Hospital.

DETAILED DESCRIPTION:
ANCA (anti-neutrophil cytoplasmic antibody)-associated vasculitis is characterised by small vessel vasculitis and presence of autoantibodies, ANCA. It can be a life-threatening disease with renal/respiratory failure. Current standard therapy in induction remission for ANCA-associated vasculitis is combination of high-dose glucocorticoid and IV-cyclophosphamide. This regimen is effective (remission rate; 80-90%), but often cause various glucocorticoid-related side effects. Especially, infection is related to death. Thus a new regimen reducing glucocorticoid dose is required.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent by a patient or a surrogate decision maker
2. Age=>20 years
3. New clinical diagnosis of ANCA-associated vasculitis (granulomatosis with polyangiitis, microscopic polyangiitis or renal limited ANCA-associated vasculitis) consistent with the 2012 Chapel Hill consensus definitions
4. Positive test by ELISA for proteinase 3-ANCA or myeloperoxidase-ANCA

Exclusion Criteria:

1. Prior treatment for ANCA-associated vasculitis before trial entry
2. ANCA-associated vasculitis related glomerulonephritis (eGFR<15ml/min) or alveolar hemorrhage (oxygen inhalation >2L/min)
3. Presence of another multisystem autoimmune disease
4. Known infection with HIV; a past or current history of hepatitis B virus or hepatitis C virus infection
5. Desire to bear children, pregnancy or lactating
6. History of malignancy within the past 5 years or any evidence of persistent malignancy
7. Ongoing or recent (last 1 year) evidence of active tuberculosis
8. Severe allergy or anaphylaxis to monoclonal antibody therapy
9. Any concomitant condition anticipated to likely require oral systemic glucocorticoids, immunosuppressants, biologics, plasma exchange or IVIg
10. Any biological B cell depleting agent (such as rituximab or belimumab) within the past 6 months
11. Other conditions, in the investigator's opinion, inappropriate for the trial entry

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of the patients achieving remission | 6 months
  Remission; BVAS ver.3=0 (or 1 with only one minor and persistent BVAS item) and prednisolone <10mg/day

SECONDARY OUTCOMES:
Time to remission | assessed at 1, 2, 4 and 6 months
  Remission; BVAS ver.3=0 (or 1 with only one minor and persistent BVAS item) and prednisolone <10mg/day
Overall survival, disease free survival, time to end-stage renal disease, time to the first serious adverse event | 0-24 months
  Assessed by Kaplan-Meier curves
Proportions of death, relapse, end-stage renal disease and the composite of these | at 6 and 24 months
  Assessed by Kaplan-Meier curves
Proportions of major relapse | at 24 months
  major relapse is relapse with one or more BVAS major items
Birmingham Vasculitis Activity Score (BVAS) version 3 | assessed at 0, 1, 2, 4, 6, 9, 12, 18 and 24 months
  BVAS is a scoring system for assessing disease activity of vasculitis
Vasculitis Damage Index (VDI) | assessed at 0, 6, 12, 18 and 24 months
  VDI is a scoring system for assessing irreversible disease damage due to vasculitis
Short-Form 36 (SF-36) | assessed at 0, 6, 12, 18 and 24 months
  SF-36 is a scoring system for assessing patient QOL.
Patient global assessment (visualised analogue scale) | assessed at 0, 6, 12, 18 and 24 months
  global assessments for disease activity and treatment toxicity
Accumulative dose of glucocorticoids | assessed at 6 and 24 months
  Accumulative dose of glucocorticoids during the study period
Numbers of events of adverse events/serious adverse events, proportions of the patients with adverse events/serious adverse events | at 6 and 24 months
  Event numbers and proportion of the patients with one or more events are assessed.
Proportions of the patients with new onset diabetes mellitus | at 6 and 24 months
  diabetes mellitus requiring drug treatments
Proportion of the patients with new onset insomnia | at 6 and 24 months
  insomnia requiring drug treatments
Proportion of the patients with new onset bone fracture, bone density | at 6 and 24 months
  bone density is assessed at lumber spines
Number of infections, proportions of the patients with infection | at 6 and 24 months
  infections requiring drug treatments
Proportions of the patients with new onset hypertension | at 6 and 24 months
  hypertension requiring drug treatments
Proportions of the patients with new onset hyperlipidemia | at 6 and 24 months
  hyperlipidemia requiring drug treatments
Proportions of patients achieving remission and discontinuance of glucocorticoids | at 6 and 24 months
  Remission is BVAS ver3=0 and prednisolone <10mg/day.

OTHER OUTCOMES:
Serum immunoglobulin levels | assessed at 0, 1, 2, 4, 6, 9, 12, 18 and 24 months
  Serum immunoglobulin levels
Peripheral blood B cell counts | assessed at 0, 1, 2, 4, 6, 9, 12, 18 and 24 months
  CD19 positive B cells assessed by FACS
serum MPO-/PR3-ANCA levels measured by ELISA | assessed at 0, 1, 2, 4, 6, 9, 12, 18 and 24 months
  MPO-ANCA and PR3-ANCA are disease specific autoantibodies binding neutrophil cytoplasmic antigen.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Nakajima, M.D., Ph.D, Principal Investigator — Chiba University Hospital
Locations (17):
- Japan (17):
  - Asahi General Hospital, Asahi, Chiba
  - Kameda Medical Centre, Kamogawa, Chiba
  - Matsudo City Hospital, Matsudo, Chiba
  - Japanese Red Cross Narita Hospital, Narita, Chiba
  - Shimoshizu Hospital, Yotsukaidō, Chiba
  - Hokkaido University, Sapporo, Hokkaido
  - Yokohama Rosai Hospital, Yokohama, Kanagawa
  - Saitama Medical Center, Kawagoe, Saitama
  - Dokkyo Medical University, Mibu, Tochigi
  - Keio University Hospital, Shinanomachi, Tokyo
  - Teikyo University, tabashi City, Tokyo
  - Akita University, Akita
  - Chiba University Hospital, Chiba
  - Chiba Aoba Municipal Hospital, Chiba
  - Chiba East Hospital, Chiba
  - Fukushima Medical University, Fukushima
  - Niigata University, Niigata

REFERENCES:
- [Background] Booth AD, Almond MK, Burns A, Ellis P, Gaskin G, Neild GH, Plaisance M, Pusey CD, Jayne DR; Pan-Thames Renal Research Group. Outcome of ANCA-associated renal vasculitis: a 5-year retrospective study. Am J Kidney Dis. 2003 Apr;41(4):776-84. doi: 10.1016/s0272-6386(03)00025-8. PMID 12666064
- [Background] de Groot K, Harper L, Jayne DR, Flores Suarez LF, Gregorini G, Gross WL, Luqmani R, Pusey CD, Rasmussen N, Sinico RA, Tesar V, Vanhille P, Westman K, Savage CO; EUVAS (European Vasculitis Study Group). Pulse versus daily oral cyclophosphamide for induction of remission in antineutrophil cytoplasmic antibody-associated vasculitis: a randomized trial. Ann Intern Med. 2009 May 19;150(10):670-80. doi: 10.7326/0003-4819-150-10-200905190-00004. PMID 19451574
- [Background] De Groot K, Rasmussen N, Bacon PA, Tervaert JW, Feighery C, Gregorini G, Gross WL, Luqmani R, Jayne DR. Randomized trial of cyclophosphamide versus methotrexate for induction of remission in early systemic antineutrophil cytoplasmic antibody-associated vasculitis. Arthritis Rheum. 2005 Aug;52(8):2461-9. doi: 10.1002/art.21142. PMID 16052573
- [Background] Jayne DR, Gaskin G, Rasmussen N, Abramowicz D, Ferrario F, Guillevin L, Mirapeix E, Savage CO, Sinico RA, Stegeman CA, Westman KW, van der Woude FJ, de Lind van Wijngaarden RA, Pusey CD; European Vasculitis Study Group. Randomized trial of plasma exchange or high-dosage methylprednisolone as adjunctive therapy for severe renal vasculitis. J Am Soc Nephrol. 2007 Jul;18(7):2180-8. doi: 10.1681/ASN.2007010090. Epub 2007 Jun 20. PMID 17582159
- [Background] Fauci AS, Wolff SM, Johnson JS. Effect of cyclophosphamide upon the immune response in Wegener's granulomatosis. N Engl J Med. 1971 Dec 30;285(27):1493-6. doi: 10.1056/NEJM197112302852701. No abstract available. PMID 5127139
- [Background] Popa ER, Stegeman CA, Bos NA, Kallenberg CG, Tervaert JW. Differential B- and T-cell activation in Wegener's granulomatosis. J Allergy Clin Immunol. 1999 May;103(5 Pt 1):885-94. doi: 10.1016/s0091-6749(99)70434-3. PMID 10329824
- [Background] Stone JH, Merkel PA, Spiera R, Seo P, Langford CA, Hoffman GS, Kallenberg CG, St Clair EW, Turkiewicz A, Tchao NK, Webber L, Ding L, Sejismundo LP, Mieras K, Weitzenkamp D, Ikle D, Seyfert-Margolis V, Mueller M, Brunetta P, Allen NB, Fervenza FC, Geetha D, Keogh KA, Kissin EY, Monach PA, Peikert T, Stegeman C, Ytterberg SR, Specks U; RAVE-ITN Research Group. Rituximab versus cyclophosphamide for ANCA-associated vasculitis. N Engl J Med. 2010 Jul 15;363(3):221-32. doi: 10.1056/NEJMoa0909905. PMID 20647199
- [Background] Jones RB, Tervaert JW, Hauser T, Luqmani R, Morgan MD, Peh CA, Savage CO, Segelmark M, Tesar V, van Paassen P, Walsh D, Walsh M, Westman K, Jayne DR; European Vasculitis Study Group. Rituximab versus cyclophosphamide in ANCA-associated renal vasculitis. N Engl J Med. 2010 Jul 15;363(3):211-20. doi: 10.1056/NEJMoa0909169. PMID 20647198
- [Background] Buch MH, Smolen JS, Betteridge N, Breedveld FC, Burmester G, Dorner T, Ferraccioli G, Gottenberg JE, Isaacs J, Kvien TK, Mariette X, Martin-Mola E, Pavelka K, Tak PP, van der Heijde D, van Vollenhoven RF, Emery P; Rituximab Consensus Expert Committee. Updated consensus statement on the use of rituximab in patients with rheumatoid arthritis. Ann Rheum Dis. 2011 Jun;70(6):909-20. doi: 10.1136/ard.2010.144998. Epub 2011 Mar 6. PMID 21378402
- [Background] Rafailidis PI, Kakisi OK, Vardakas K, Falagas ME. Infectious complications of monoclonal antibodies used in cancer therapy: a systematic review of the evidence from randomized controlled trials. Cancer. 2007 Jun 1;109(11):2182-9. doi: 10.1002/cncr.22666. PMID 17429839
- [Background] Walsh M, Merkel PA, Mahr A, Jayne D. Effects of duration of glucocorticoid therapy on relapse rate in antineutrophil cytoplasmic antibody-associated vasculitis: A meta-analysis. Arthritis Care Res (Hoboken). 2010 Aug;62(8):1166-73. doi: 10.1002/acr.20176. PMID 20235186
- [Background] Wada T, Hara A, Arimura Y, Sada KE, Makino H; Research Group of Intractable Vasculitis, Ministry of Health, Labor, and Welfare of Japan. Risk factors associated with relapse in Japanese patients with microscopic polyangiitis. J Rheumatol. 2012 Mar;39(3):545-51. doi: 10.3899/jrheum.110705. Epub 2011 Dec 15. PMID 22174198
- [Background] Furuta S, Chaudhry AN, Hamano Y, Fujimoto S, Nagafuchi H, Makino H, Matsuo S, Ozaki S, Endo T, Muso E, Ito C, Kusano E, Yamagata M, Ikeda K, Kashiwakuma D, Iwamoto I, Westman K, Jayne D. Comparison of phenotype and outcome in microscopic polyangiitis between Europe and Japan. J Rheumatol. 2014 Feb;41(2):325-33. doi: 10.3899/jrheum.130602. Epub 2014 Jan 15. PMID 24429174
- [Background] Smith RM, Jones RB, Guerry MJ, Laurino S, Catapano F, Chaudhry A, Smith KG, Jayne DR. Rituximab for remission maintenance in relapsing antineutrophil cytoplasmic antibody-associated vasculitis. Arthritis Rheum. 2012 Nov;64(11):3760-9. doi: 10.1002/art.34583. PMID 22729997
- [Background] Jennette JC, Falk RJ, Bacon PA, Basu N, Cid MC, Ferrario F, Flores-Suarez LF, Gross WL, Guillevin L, Hagen EC, Hoffman GS, Jayne DR, Kallenberg CG, Lamprecht P, Langford CA, Luqmani RA, Mahr AD, Matteson EL, Merkel PA, Ozen S, Pusey CD, Rasmussen N, Rees AJ, Scott DG, Specks U, Stone JH, Takahashi K, Watts RA. 2012 revised International Chapel Hill Consensus Conference Nomenclature of Vasculitides. Arthritis Rheum. 2013 Jan;65(1):1-11. doi: 10.1002/art.37715. No abstract available. PMID 23045170
- [Background] Exley AR, Bacon PA, Luqmani RA, Kitas GD, Gordon C, Savage CO, Adu D. Development and initial validation of the Vasculitis Damage Index for the standardized clinical assessment of damage in the systemic vasculitides. Arthritis Rheum. 1997 Feb;40(2):371-80. doi: 10.1002/art.1780400222. PMID 9041949
- [Derived] Furuta S, Nakagomi D, Kobayashi Y, Hiraguri M, Sugiyama T, Amano K, Umibe T, Kono H, Kurasawa K, Kita Y, Matsumura R, Kaneko Y, Ninagawa K, Hiromura K, Kagami SI, Inaba Y, Hanaoka H, Ikeda K, Nakajima H; LoVAS collaborators. Reduced-dose versus high-dose glucocorticoids added to rituximab on remission induction in ANCA-associated vasculitis: predefined 2-year follow-up study. Ann Rheum Dis. 2024 Jan 2;83(1):96-102. doi: 10.1136/ard-2023-224343. PMID 37734880
- [Derived] Furuta S, Nakagomi D, Kobayashi Y, Hiraguri M, Sugiyama T, Amano K, Umibe T, Kono H, Kurasawa K, Kita Y, Matsumura R, Kaneko Y, Ninagawa K, Hiromura K, Kagami SI, Inaba Y, Hanaoka H, Ikeda K, Nakajima H; LoVAS Collaborators. Effect of Reduced-Dose vs High-Dose Glucocorticoids Added to Rituximab on Remission Induction in ANCA-Associated Vasculitis: A Randomized Clinical Trial. JAMA. 2021 Jun 1;325(21):2178-2187. doi: 10.1001/jama.2021.6615. PMID 34061144
- [Derived] Serling-Boyd N, Wallace ZS. Management of primary vasculitides with biologic and novel small molecule medications. Curr Opin Rheumatol. 2021 Jan;33(1):8-14. doi: 10.1097/BOR.0000000000000756. PMID 33164993
- [Derived] Furuta S, Sugiyama T, Umibe T, Kaneko Y, Amano K, Kurasawa K, Nakagomi D, Hiraguri M, Hanaoka H, Sato Y, Ikeda K, Nakajima H; LoVAS Trial study investigators. Low-dose glucocorticoids plus rituximab versus high-dose glucocorticoids plus rituximab for remission induction in ANCA-associated vasculitis (LoVAS): protocol for a multicentre, open-label, randomised controlled trial. BMJ Open. 2017 Dec 14;7(12):e018748. doi: 10.1136/bmjopen-2017-018748. PMID 29247107